CLINICAL TRIAL: NCT01601314
Title: Perioperative Magnesium Sulphate as a Cerebral Protector in Neurosurgical Patients
Acronym: MAGNA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sara Varea (Other)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MAGNA; 2011-006301-10 (EudraCT Number)
Record Dates: First submitted 2012-05-10; First posted 2012-05-18 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Seizures (Incl Subtypes); Brain Tumor
MeSH Terms: conditions — Seizures; Brain Neoplasms | interventions — Magnesium Sulfate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- magnesium sulphate (Experimental): The patients who are going to receive Magnesium Sulphate
  Interventions: Drug: Magnesium Sulfate
- Control (Placebo Comparator): Patients who are going to receive Sodium Chloride 0.9%
  Interventions: Other: Sodium Chloride

INTERVENTIONS:
Drug: Magnesium Sulfate — At the beginning of the neurosurgery, the subjects are going to receive one 4gr bolus in Sodium Chloride 100 mL, lasting 20 minutes, intravenously.
  After that, a intravenously perfusion of Magnesium Sulfate 20 gr, in Sodium Chloride 1000 mL, lasting 24 hours, will be started.
  Arms: magnesium sulphate
Other: Sodium Chloride — At the beginning of the neurosurgery, the subjects are going to receive a bolus of Sodium Chloride 100 mL, lasting 20 minutes, intravenously.
  After that, a intravenously perfusion of Sodium Chloride 1000 mL, lasting 24 hours, will be started.
  Arms: Control

SUMMARY:
The purpose of this study is to determine the relationship between magnesium sulphate administration and levels of S100B protein in serum of patients undergoing supratentorial brain parenchymal resection.

ELIGIBILITY:
Inclusion Criteria:

* Male and females older than 18 years.
* Undergoing supratentorial parenchyma resection surgery.
* Capable of collaborate on probes and explorations included in the study.
* Signature the written informed consent form.

Exclusion Criteria:

* Life expectancy less than 12 months due to the suspected histological type of tumour.
* Hypothalamic-pituitary axis illness.
* Presence of Melanoma previously.
* Glomerular filtration rate less than 60 mL/min.
* Thyroid or parathyroid glands pathology.
* Myasthenia gravis.
* Respiratory depression.
* Pregnancy or breastfeeding.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum S100B protein | 2 hours after the end of the surgery

SECONDARY OUTCOMES:
Serum S100B protein | 1 hour before surgery; daily postoperative until day 10.
Serum Specific Neuronal Enolase (SNE) | 1 hour before surgery; 2 hours after end of surgery; every 48 hours until day 10
Improvement on Magnetic Resonance Imaging | within the month prior to surgery; early postoperative; 6 months postoperative
Improvement on Neuropsychological Assessment | within the month prior to surgery; early postoperative; 1, 6 and 12 months postoperative
Glasgow Outcome Scale | 6 and 12 month postoperative
Mortality | 6 and 12 month postoperative
Apolipoprotein E genotype | 1 hour before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Neus Fabregas, MD PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clinic of Barcelona, Barcelona, Spain